CLINICAL TRIAL: NCT02903134
Title: Early Risk of Asthma in Children Exposed to In-utero Maternal Obesity: An Epigenetic-mediated Programming of Immune Function
Brief Title: Early Risk of Asthma in Children Exposed to In-utero Maternal Obesity
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 13-225; FONDECYT 1141195 (Other Grant/Funding Number: CONICYT-FONDECYT)
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2018-06

CONDITIONS: Asthma; Children; Obesity; Maternal
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood sample, cord blood sample and skin prick test.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborn from obese and nonobese pregnant: Obese (BMI>30) or normal weight (BMI<25) women at their first antenatal visit were invited to participate in the study at the moment of delivery at Sotero del Rio Hospital, Santiago. Information regarding birth outcomes, parental history, as well as environmental conditions was collected at recruitment. Follow-up questionnaires by phone were completed every 6 months. Umbilical cord blood samples were collected to measure IL-12, TNF-α, IL-10, IL-4; to evaluate metabolic status; to isolated monocytes and macrophage differentiation; and for DNA methylation status of the promoter regions of the genes coding for TNF-α, IL-12, IL-10, and IL-4Rα. Also, fasting blood samples of the mothers within 48 hours after delivery; and blood samples and skin prick test were collected.

SUMMARY:
This study seeks a better understanding of the pathogenesis of asthma in early life. The aim of this project is to determine whether the offspring of obese mothers at 3 years of life have increased the risk of asthma compared to children whose mothers were not obese and whether this increased risk is associated with a programming altered immune reactivity at birth.

DETAILED DESCRIPTION:
The general objectives of this study are:

1. To determine whether the increased risk of asthma in children born from a pre-pregnant obese mother can be observed at 3 years of life and whether this increased risk associated with altered plasma levels of immune mediators at birth.
2. To explore in children born from pre-pregnant obese mother whether monocyte physiology and M1-M2 polarization present an altered response and expression of asthma-related immune-modulations at birth.
3. To study in neonates born from pre-pregnant obese mother whether the in vitro expression of TNFα, IL12, IL-10 and IL-4Rα in monocytes associates with changes in the DNA methylation status in the promoter regions of those genes.

The study is performed in accordance with the Helsinki Declaration, and the study protocol was accepted by Institutional Review Boards at School of Medicine of the Pontificia Universidad Católica de Chile.

ELIGIBILITY:
Inclusion Criteria:

* Women who receive care in any of the 12 public health care centers in La Florida and Puente Alto and give birth in the Sotero del Río Hospital.
* Singleton pregnancy of fewer than 14 weeks of gestation at the first antenatal visit.
* 18 years or older

Exclusion Criteria:

* Pregnant women with overweight (BMI 25-30) before 14 weeks.
* Women that have a premature birth, cardio-respiratory disorder or neurological defects of the neonate.
* Women that develop gestational diabetes and hypertension during pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The recruitment of participants was performed in the Sotero del Rio Hospital at Santiago. Women that were obese (BMI>30) or normal weight (BMI<25) at their first antenatal visit were invited to participate in the study at the moment of delivery.
  Questionnaires: Information regarding birth outcomes, maternal and paternal history of asthma and allergy, as well as environmental conditions at home (pet ownership, indoor smoking, heating system, and so on) was collected using a questionnaire at the moment of recruitment.
  Follow-up questionnaires by phone are completed every 6 months. These questionnaires collect information regarding diagnosis of asthma/allergy and acute respiratory illness, environmental conditions, and relevant confounding variables
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Risk of asthma (defined as "positive asthma predictive index" at 36 months of age) | 36 months of age

SECONDARY OUTCOMES:
Allergy status (positive skin prick test) | 30-36 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Castro-Rodriguez, MD, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castro-Rodriguez JA, Forno E, Casanello P, Padilla O, Krause BJ, Uauy R. Leptin in Cord Blood Associates with Asthma Risk at Age 3 in the Offspring of Women with Gestational Obesity. Ann Am Thorac Soc. 2020 Dec;17(12):1583-1589. doi: 10.1513/AnnalsATS.202001-080OC. PMID 32726560
- [Result] Cifuentes-Zuniga F, Arroyo-Jousse V, Soto-Carrasco G, Casanello P, Uauy R, Krause BJ, Castro-Rodriguez JA. IL-10 expression in macrophages from neonates born from obese mothers is suppressed by IL-4 and LPS/INFgamma. J Cell Physiol. 2017 Dec;232(12):3693-3701. doi: 10.1002/jcp.25845. Epub 2017 Apr 27. PMID 28160500
- [Result] Vega-Tapia F, Artigas R, Hernandez C, Uauy R, Casanello P, Krause BJ, Castro-Rodriguez JA. Maternal obesity is associated with a sex-specific epigenetic programming in human neonatal monocytes. Epigenomics. 2020 Nov;12(22):1999-2018. doi: 10.2217/epi-2020-0098. Epub 2020 Dec 4. PMID 33275450
- [Result] Jaramillo-Ospina A, Castano-Moreno E, Munoz-Munoz E, Krause BJ, Uauy R, Casanello P, Castro-Rodriguez JA. Maternal Obesity Is Associated With Higher Cord Blood Adipokines in Offspring Most Notably in Females. J Pediatr Gastroenterol Nutr. 2021 Aug 1;73(2):264-270. doi: 10.1097/MPG.0000000000003172. PMID 34016877
- [Result] Castro-Rodriguez JA, Forno E, Padilla O, Casanello P, Krause BJ, Borzutzky A. The asthma predictive index as a surrogate diagnostic tool in preschoolers: Analysis of a longitudinal birth cohort. Pediatr Pulmonol. 2021 Oct;56(10):3183-3188. doi: 10.1002/ppul.25592. Epub 2021 Jul 28. PMID 34320686